CLINICAL TRIAL: NCT01725659
Title: Innovative Modalities for Restoring Upper Limb Function Post Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malcom Randall VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Janis Daly, Principal Investigator, Malcom Randall VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2801R
Record Dates: First submitted 2012-11-09; First posted 2012-11-14 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Cerebrovascular Accident
Keywords: Stroke; electric stimulation; robotics; motor learning
MeSH Terms: conditions — Stroke | interventions — Robotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Motor Learning (Experimental): subjects are provided with intensive motor learning training of the upper limb
  Interventions: Other: Motor Learning
- Robotics and Motor Learning (Experimental): subject are provided with intensive motor learning and robotics training of the upper limb
  Interventions: Other: Motor Learning; Other: Robotics
- Motor learning and FES (Experimental): subjects are provided with intensive motor learning and surface FES (Functional Electrical Stimulation) of the upper limb
  Interventions: Other: Motor Learning; Other: surface FES

INTERVENTIONS:
Other: Motor Learning — training of the hemiplegic upper limb with motor learning
Other: Robotics — subjects perform training of hemiplegic arm using an upper extremity robot
  Arms: Robotics and Motor Learning
Other: surface FES — subjects are provided with surface FES to the hemiplegic upper limb
  Arms: Motor learning and FES

SUMMARY:
PURPOSE. After stroke many patients are unable to engage in normal upper limb functional activities, which may restrict them from participation in meaningful life roles. For many, conventional rehabilitation does not restore upper limb function to a useful level. The purpose of this research is to investigate the benefits of three promising motor learning interventions: focused intensive, motor learning (FIML); 2) robotics and motor learning (ROB-ML); and 3) functional neuromuscular stimulation and motor learning (FNS-ML).

ELIGIBILITY:
Inclusion Criteria:

* >1 year post stroke no acute, uncontrolled medical condition single stroke

Exclusion Criteria:

* pacemaker other neurological condition more than one stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2001-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Fugl Meyer | after 12 weeks of intervention
  impairment measure of coordination of the upper limb

CONTACTS AND LOCATIONS:
Locations (1):
- Louis Stokes Cleveland Department of Veterans Affairs Medical Center, Cleveland, Ohio, United States